CLINICAL TRIAL: NCT00319969
Title: A Randomized Phase 2 Trial Comparing Amrubicin Versus Topotecan as Second-Line Treatment in Patients With Extensive Small Cell Lung Cancer Sensitive to First-Line Chemotherapy
Brief Title: Study Comparing Amrubicin Versus Topotecan in Patients With Small Cell Lung Cancer Who Have Responded to Prior Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Kathy Knapp, Clinical Program Manager, Pharmion Corporation
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNF3140-SCLC-05004
Expanded Access: Available
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; amrubicin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — amrubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Amrubicin 40mg/m<2> IV days 1, 2, 3 of each 21-day cycle until disease progression.
  Interventions: Drug: Amrubicin
- 2 (Active Comparator): Topotecan 1.5mg/m<2> IV, days 1, 2, 3, 4, 5 of each 21-day cycle until disease progression.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Amrubicin — Amrubicin 40mg/m<2> IV days 1, 2, 3 of each 21-day cycle until disease progression.
  Arms: 1
Drug: Topotecan — Topotecan 1.5mg/m<2> IV days 1, 2, 3, 4, 5 of each 21-day cycle until disease progression.
  Other Names: Hycamtin(R)
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the objective tumor response rate of amrubicin or standard topotecan therapy when administered as second-line therapy to ED-SCLC patients who have chemotherapy sensitive recurrent or progressive.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of SCLC
* Extensive disease (ED) at time of study entry
* Response to first-line platinum-based chemotherapy
* Recurrent or progressive SCLC ≥90 days after completion of first-line therapy
* At least 18 years of age
* ECOG Performance Status of 0, 1, or 2
* Measurable disease defined by RECIST criteria

  * Measurable disease: The presence of at least one measurable lesion. If only one lesion is present, the neoplastic nature of the disease site should be confirmed by histology and/or cytology.
  * Measurable lesion: Lesions that can be accurately measured in at least one dimension with the longest diameter ≥20mm using conventional techniques or ≥10mm using spiral CT scans.

CT (including spiral CT) scans and MRI are the preferred methods of measurement; however, chest x-rays are acceptable if the leions are clearly defined and surrounded by aerated lung. Clinically detected lesions will only be considered measurable when they are superficial (eg., skin nodules and palpable lymph nodes). For the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion is required.

* Adequate organ function including the following:

  * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥1500 cells/μL, platelet count ≥100,000 cells/μL and hemoglobin ≥9 g/dL
  * Hepatic: bilirubin ≤1.5 X ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 X ULN
  * Renal: serum creatinine <2.0mg/dL or calculated creatinine clearance >60mL/min
  * Cardiac: Left ventricular ejection fraction (LVEF) ≥50%
* Negative serum pregnancy test at the time of enrollment for women of child-bearing potential. For men and women of child-producing potential, use of effective contraceptive methods during the study.
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments

Exclusion Criteria:

* Pregnant or nursing women
* Chest radiotherapy within the previous 28 days or other radiotherapy within the previous 14 days. Recovery from the acute toxic effects of radiation required prior to study enrollment. Measurable lesions that have been previously irradiated must be enlarging to be considered target lesions. Prior radiation therapy allowed to <25% of the bone marrow.
* More than 1 prior chemotherapy regimen for SCLC
* Prior anthracycline treatment
* Participation in any investigational drug study within 28 days prior to study entry
* Patients with second primary malignancy (except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin or other malignancy treated at least 5 years previously with no evidence of recurrence; prior low grade [Gleason score ≤6] localized prostate cancer is allowed)
* Concurrent severe or uncontrolled medical disease (i.e., active systemic infection, diabetes, hypertension, coronary artery disease, congestive heart failure) that, in the opinion of the Investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study.
* Symptomatic central nervous system metastases. Patients with asymptomatic brain metastases are allowed. The patient must be stable after radiotherapy for ≥2 weeks and off corticosteroids for ≥1 week.
* History of interstitial lung disease or pulmonary fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate | Until Disease Progression

SECONDARY OUTCOMES:
Time to tumor progression | Until Disease Progression
Progression free survival | Until death or disease progression
Overall survival (median survival time; 1 year survival) | Until death
Toxicity profile | Until 30 days after final dose
Incidence of cumulative cardiomyopathy | Until end of study participation
Regression of CNS metastases | Until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Ungerleider, MD, Study Director — Theradex
Locations (47):
- United States (47):
  - Birmingham Hematology & Oncology, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Alta Bates Medical Center - Comprehensive Cancer Center, Berkeley, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Rocky Mountain Cancer Center - Denver, Denver, Colorado
  - Rocky Mountain Cancer Center - Sky Ridge, Lone Tree, Colorado
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, PA, Ocoee, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Cancer Care & Hematology Specialists of Chicago, Niles, Illinois
  - Oncology & Hematology of Central Illinois, Peoria, Illinois
  - Blessing Cancer Center, Quincy, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Hope Center, Terre Haute, Indiana
  - Norton Healthcare - Louisville Oncology, Louisville, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins Hospital - The Bunting Blaustein Cancer Research Building, Baltimore, Maryland
  - Maryland Oncology Hematology, PA, Columbia, Maryland
  - Alliance Hematology Oncology, PA - Carroll County Cancer Center, Westminster, Maryland
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Hematology/Oncology Consultants, St Louis, Missouri
  - Arch Medical Services - Center for Cancer Care & Research, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology, PC, Albany, New York
  - SUNY Upstate Medical University - Regional Oncology Center, Syracuse, New York
  - Northwestern Carolina Oncology & Hematology, Hickory, North Carolina
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Northwest Cancer Specialists, Portland, Oregon
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, PA, Dallas, Texas
  - Texas Oncology - Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, PA, Fort Worth, Texas
  - Alison Cancer Center, Midland, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care & Research Center, Waco, Texas
  - Texas Oncology, PA - Deke Slayton Cancer Center, Webster, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology & Hematology Associates of SW Virginia, Inc., Salem, Virginia
  - Puget Sound Cancer Center, Seattle, Washington
  - Northwest Cancer Specialists - Vancouver Cancer Center, Vancouver, Washington